CLINICAL TRIAL: NCT06145100
Title: Evaluation of Ultrasound Parameters and Liver and Spleen Stiffness for Prediction of Clinically Significant Portal Hypertension in Patients With Common Variable Immunodeficiency Syndrome
Brief Title: Prediction of Portal Hypertension in Patients With CVID (CVID-pHT)
Acronym: CVID-pHT
Status: Recruiting | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dominik Bettinger, Principal Investigator, University Hospital Freiburg
Other Study IDs: CVID-pHT
Record Dates: First submitted 2023-11-10; First posted 2023-11-22 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Non-Cirrhotic Portal Hypertension; Common Variable Immunodeficiency
Keywords: non-cirrhotic portal hypertension; Common Variable Immunodeficiency; ultrasound; liver stiffness measurement; spleen stiffness measurement
MeSH Terms: conditions — Common Variable Immunodeficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, peripheral blood mononuclear cell (PBMC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with CVID and autoimmunity and no liver involvement.: Patients with CVID and autoimmune disease, but no liver involvement (normal liver enzymes and normal abdominal ultrasound)
  Interventions: Diagnostic Test: Ultrasound including color doppler ultrasound
- Patients with CVID and liver involvement and no clinical significant portal hypertension: Patients with CVID and liver involvement (elevated liver enzymes, abnormal ultrasound and/or abnormal liver biopsy), but no clinically significant portal hypertension
  Interventions: Diagnostic Test: Ultrasound including color doppler ultrasound
- Patients with CVID and clinically significant non-cirrhotic portal hypertension: Patients with CVID and clinically significant non-cirrhotic portal hypertension (indicated by the presence of ascites or esophageal varices / portal-hypertensive gastropathy).
  Interventions: Diagnostic Test: Ultrasound including color doppler ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound including color doppler ultrasound — Patients with CVID receive color doppler ultrasound of the liver including assessment of portal vein diameter, portal vein flow velocity, hepatic vein diameter and assessment of arterial perfusion. Further liver and spleen stiffness measurement by transient elastography is performed.
  Other Names: Liver stiffness measurement by transient elastography; Spleen stiffness measurement by transient elastography

SUMMARY:
Patients with CVID will be offered to participate in this observational trial during the routine annual visit in the outpatient clinic at the Center of chronic Immunodeficiency (CCI) of the University Medical Center Freiburg, Germany.

Clinical and laboratory data at the time of presentation will be assessed. Additionally, parameters of abdominal ultrasound, duplex sonography of the liver and spleen, and liver and spleen stiffness at the time of presentation will be evaluated. If applicable, clinical and/or interventional parameters indicating clinically significant portal hypertension (i.e. presence of varices or portal-hypertensive gastropathy in esophago-gastroduodenoscopy, presence of ascites) within 12 months prior and after the index visit will be assessed. During the visit, serum/plasma samples and peripheral blood mononuclear cells (PBMC) are collected and stored in an associated biobank.

DETAILED DESCRIPTION:
Patients with CVID can be included in the study. The study cohort will consist of three subgroups: 1) Patients with CVID and autoimmunity, but no liver involvement. 2) Patients with CVID and liver involvement, defined by elevated liver enzymes, abnormal ultrasound and/or abnormal liver biopsy, but no signs of clinically significant portal hypertension and 3) Patients with CVID and clinically significant non-cirrhotic portal hypertension. Further, patients with CVID and diagnosed non-cirrhotic portal hypertension between 01/01/2004 and the start of the prospective part of this study (01/01/2023) will be included retrospectively in this study.

Patients will be recruited during the routine annual visit in the outpatient clinic at the Center of chronic Immunodeficiency (CCI) of the University Medical Center Freiburg, Germany. During the visit a standard ultrasound protocol, including size and morphology of liver and spleen, duplex-sonography of the liver, and measurement of liver and spleen stiffness via transient elastography will be performed as a part of the routine clinical diagnostic. Results from endoscopy or other interventions (esophago-gastroduodenoscopy, invasive measurement of hepatic venous-portal pressure gradient, or TIPS implantation, if applicable) within 12 months prior and after the index visit will be assessed. All non-invasive and invasive interventions will be conducted solely based on clinical decisions made independently from the study inclusion as the study is designed as an observational study.

Detailed patient characteristics, epidemiologic, clinical, imaging and laboratory parameters will be assessed and included in an electronic database.

Apart from these data, patients will be asked to participate in biobank sampling including serum/plasma and peripheral blood mononuclear cells (PBMC) samples from the peripheral veins.

All patients recruited in this study will be followed-up for at least 12 months.

Outcome parameters include parameters from abdominal ultrasound, duplex-sonography and stiffness of liver and spleen, presence or development of clinically significant portal hypertension and non-invasive fibrosis scores based on laboratory and ultrasound parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CVID

Exclusion Criteria:

* no written informed consent
* concomitant chronic liver disease (viral hepatitis, alcoholic liver disease, steatitic liver disease, hemochromatosis, primary biliary cholangitis, primary sclerosis cholangitis, M. Wilson, alpha-1-antitrypsin deficiency)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CVID will be included in the study. Patients will be divided into three subgroups: 1) Patients with CVID and autoimmunity, but no liver involvement (n=75) 2) Patients with CVID and liver involvement, defined by elevated liver enzymes, abnormal ultrasound and/or abnormal liver biopsy, but no signs of clinically significant portal hypertension (n=75) 3) Patients with CVID and clinically significant non-cirrhotic portal hypertension (n=75).
  Further patients with CVID and diagnosed non-cirrhotic portal hypertension between 01/01/2004 and the start of the prospective part of this study (01/01/2023) will be included retrospectively in this study (n=25)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in liver stiffness between CVID patients with and without liver involvement and with clinically significant portal hypertension. | Study inclusion, after 12 months
  Liver stiffness will be assessed by transient elastography.
Differences in spleen stiffness between CVID patients with and without liver involvement and with clinically significant portal hypertension. | Study inclusion, after 12 months
  Spleen stiffness will be assessed by transient elastography.

SECONDARY OUTCOMES:
Differences in portal vein diameter between CVID patients with and without liver involvement and with clinically significant portal hypertension. | Study inclusion, after 12 months
  Portal vein diameter will be assessed by color doppler ultrasound
Differences in portal vein flow velocity between CVID patients with and without liver involvement and with clinically significant portal hypertension. | Study inclusion, after 12 months
  Portal vein flow velocity will be assessed by color doppler ultrasound
Differences in alanine aminotransfersases (ALT) between CVID patients with and without liver involvement and with clinically significant portal hypertension. | Study inclusion, after 12 months
  ALT is assessed during routine clinical practice
Differences in aspartat aminotransfersases (AST) between CVID patients with and without liver involvement and with clinically significant portal hypertension. | Study inclusion, after 12 months
  AST is assessed during routine clinical practice
Differences in liver function tests (bilirubin, albumin, INR) between CVID patients with and without liver involvement and with clinically significant portal hypertension. | Study inclusion, after 12 months
  Liver function liver function tests (bilirubin, albumin, INR) are assessed during routine clinical practice
Differences in platelets between CVID patients with and without liver involvement and with clinically significant portal hypertension. | Study inclusion, after 12 months
  Platelets are assessed during routine clinical practice

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Bettinger, MD, Principal Investigator — University Hospital Freiburg; Klaus Warnatz, MD, Principal Investigator — University Hospital Freiburg; Marlene Reincke, MD, Principal Investigator — University Hospital Freiburg
Locations (1):
- University Medical Center Freiburg, Department of Medicine II, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: Undecided